CLINICAL TRIAL: NCT04235205
Title: Efficacy and Safety of Elobixibat in Combination With Cholestyramine for Patients With Nonalcoholic Fatty Liver Disease: a Single Center, Double-blind, Randomized, Placebo-Controlled, Phase 2a Trial.
Brief Title: Efficacy and Safety of Elobixibat in Combination With Cholestyramine for Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yokohama City University (Other)
Collaborators: EA Pharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Takaomi Kessoku, Department of palliative care center, Yokohama City University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YCU19002
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
Keywords: Elobixibat; Cholestyramine; Nonalcoholic fatty liver disease; Nonalcoholic steatohepatitis; phase 2 trial; Combination therapy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — elobixibat; Cholestyramine Resin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Elobixibat and cholestyramine (Experimental): The investigational product per dosing (elobixibat 10mg and cholestyramine powder 9g) are orally administered once daily for 16 weeks.
  Interventions: Drug: Elobixibat 10mg + cholestyramine powder 9g (cholestyramine 4g)
- Elobixibat (Experimental): The investigational product per dosing (elobixibat 10mg and cholestyramine powder placebo) are orally administered once daily for 16 weeks.
  Interventions: Drug: Elobixibat 10mg + cholestyramine powder placebo
- cholestyramine (Experimental): The investigational product per dosing (elobixibat placebo and cholestyramine powder 9g) are orally administered once daily for 16 weeks.
  Interventions: Drug: Elobixibat placebo + cholestyramine powder 9g (cholestyramine 4g)
- Placebo (Placebo Comparator): The investigational product per dosing (elobixibat placebo and cholestyramine powder placebo) are orally administered once daily for 16 weeks.
  Interventions: Drug: Elobixibat placebo + cholestyramine powder placebo

INTERVENTIONS:
Drug: Elobixibat 10mg + cholestyramine powder 9g (cholestyramine 4g) — Patients with nonalcoholic fatty liver disease are administered Elobixibat 10mg + cholestyramine powder 9g (cholestyramine 4g) for 16 weeks
  Other Names: AJG533 10 mg + CTM27 9 g
  Arms: Elobixibat and cholestyramine
Drug: Elobixibat 10mg + cholestyramine powder placebo — Patients with nonalcoholic fatty liver disease are administered Elobixibat 10mg+ cholestyramine powder placebo for 16 weeks
  Other Names: AJG533 10 mg + CTM27 placebo
  Arms: Elobixibat
Drug: Elobixibat placebo + cholestyramine powder 9g (cholestyramine 4g) — Patients with nonalcoholic fatty liver disease are administered Elobixibat placebo+ cholestyramine powder 9g (cholestyramine 4g) for 16 weeks
  Other Names: AJG533 placebo + CTM27 9g
  Arms: cholestyramine
Drug: Elobixibat placebo + cholestyramine powder placebo — Patients with nonalcoholic fatty liver disease are administered Elobixibat placebo+ cholestyramine powder placebo for 16 weeks
  Other Names: AJG533 placebo + CTM27 placebo
  Arms: Placebo

SUMMARY:
The objective is to evaluate the efficacy and safety of once-daily oral doses of 10 mg elobixibat in combination with 9g cholestyramine powder (cholestyramine 4g) in patients with nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
This is a placebo-controlled, randomized, double-blind, parallel group, comparative study, when patients with nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH), are administered elobixibat at 10 mg and cholestyramine powder at 9g( cholestyramine 4g) once daily for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received adequate explanation about this study and provided written informed consent
* Patients who are ≥ 20 and < 75 years of age at the time of informed consent
* Patients who have a current biopsy-confirmed NASH within 8 months of screening or a suspected diagnosis of NAFLD/NASH based on the criteria outlined below:

  1. Biopsy-confirmed NASH is defined as histological NASH diagnosis with fibrosis stage F1 through F3 and a NAFLD activity score (NAS) of ≥4 with a score of ≥1 in each of the NAS components below as assessed by a pathologist using the NASH Clinical Research Network criteria:

     i. Steatosis (scored 0 to 3)

     ii. Ballooning degeneration (scored 0 to 2)

     iii. Lobular inflammation (scored 0 to 3)
  2. The suspected diagnosis of NAFLD/NASH is based on the following criteria:

     i. Serum aspartate aminotransferase (AST) ≥20 U/L and alanine aminotransferase (ALT) ≥40 U/L in males or ≥28 U/L in females

     ii. Waist circumference ≥85 cm in males or ≥90 cm in females

     iii. Diagnosis of metabolic syndrome having 2 or more of the following 3 risk factors at Screening:
     1. Fasting plasma glucose ≥110 mg/dL or undergoing drug treatment for elevated glucose
     2. Systolic blood pressure ≥130 mmHg and/or diastolic blood pressure≥85mmHg or undergoing drug treatment for hypertension, or antihypertensive drug treatment in a patient with a history of hypertension
     3. Triglycerides (TGs) ≥150 mg/dL or undergoing drug treatment for elevated triglycerides,and/or high-density lipoprotein-cholesterol (HDL-C)<40mg/dL or undergoing drug treatment for reduced HDL-C
* Screening Magnetic Resonance Imaging (MRI) -Proton Density Fat Fraction (PDFF) with ≥8% liver steatosis
* Fasting serum low density lipoprotein-cholesterol (LDL-C) >120 mg/dL or undergoing antidyslipidemic drugs
* Be willing to maintain a stable diet and physical activity throughout the course of the study

Exclusion criteria：

* Women who are pregnant, breastfeeding, possibly pregnant or do not agree to use birth control during the study
* Body mass index (BMI) <23 kg/m²
* Magnetic Resonance Elastography (MRE) value >6.7 kPa
* Any of the following laboratory abnormalities:

  1. ALT >5 × upper limit normal (ULN) or AST >5 × ULN
  2. Prothrombin time - international normalized ratio (PT-INR) ≥1.3 unless on anticoagulant therapy
  3. Total bilirubin > ULN, except with an established diagnosis of Gilbert's syndrome
  4. Platelet count < 80,000/μL
  5. eGFR <45 as calculated by the body surface area (BSA) adjustment (normalized eGFR)
* Acute or chronic liver disease other than NAFLD/NASH including but not limited to the following:

  1. Hepatitis B (as defined by the presence of hepatitis B surface [HBs] antigen at Screening) or hepatitis C(as defined by the presence of hepatitis C virus [HCV] antibody [anti-HCV]) Patients with positive anti-HCV who test negative for HCV ribonucleic acid (HCV-RNA) at Screening will be allowed to participate in the study as long as there is evidence of viral negativity for a minimum of 12 months prior to Screening
  2. Evidence of autoimmune hepatitis
  3. History of primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, alpha-1-anti-trypsin deficiency, hemochromatosis or iron overload, drug-induced or alcoholic liver disease, or known bile duct obstruction.
  4. Suspected or proven hepatocellular carcinoma
* Known history of human immunodeficiency virus (HIV)
* Medical history of liver cirrhosis
* Clinical evidence of portal hypertension to include any history of ascites, hepatic encephalopathy, or presence of esophageal varices
* Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines,tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, or valproic acid) or other known hepatotoxins for ≥2 weeks in the year prior to Screening
* Use of the following medications:

  1. Glucagon-like peptide-1 (GLP-1) agonists unless on a stable dose 3 months prior to Screening or liver biopsy
  2. Ursodeoxycholic acid or thiazolidinediones within 3 months prior to Screening
  3. Antidyslipidemic drugs have been stable for ≥3 months prior to Screening
  4. Oral antidiabetic drugs have been stable for ≥3 months prior to Screening
  5. Agents (including herbal over-the-counter weight loss preparations) or medications known to significantly impact body weight within 3 months prior to Screening
* History of significant alcohol consumption, defined as an average of≥20g/day in female patients and ≥30 g/day in male patients, for a period of >3 consecutive months within 1 year prior to Screening, hazardous alcohol use (Alcohol Use Disorders Identification Test score ≥8), or an inability to reliably quantify alcohol consumption but determined as alcohol polydipsia based upon judgment of the Investigator or subinvestigator
* Weight change ≥10% within the 6 months prior to Screening or ≥5% within the 3 months prior to Screening
* Surgery planned during the study period or after bariatric surgery (e.g., gastroplasty and roux-en-Y gastric bypass)
* Type 1 diabetes by medical history
* Uncontrolled Type 2 diabetes defined as hemoglobin A1c (HbA1c) >9.5% at Screening(patients with HbA1c >9.5% may be rescreened) or requiring insulin dose adjustment >10% within 2 months prior to Screening
* Clinical hyperthyroidism or hypothyroidism or Screening hormone results pointing to thyroid dysfunction. Patients receiving dose-stable thyroid replacement therapy for ≥3 months prior to Screening will be allowed to participate in this study as long as thyroid tests show that the patient is euthyroid and stable
* History of any condition causing malabsorption such as chronic pancreatitis, extensive bowel/small intestine surgery, celiac disease, or bile flow obstruction
* History of any condition associated with acute or chronic diarrhea such as inflammatory bowel disease (IBD),functional diarrhea, irritable bowel syndrome (IBS) with predominant diarrhea, IBS with mixed bowel habits, or unclassified IBS
* Uncontrolled hypertension (either treated or untreated) defined as systolic blood pressure >160 mmHg or a diastolic blood pressure >100 mmHg at Screening
* History of New York Heart Association (NYHA) Class III or IV heart failure, or known left ventricular ejection fraction <30%
* History of myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or stroke or major surgery within 6 months prior to Screening
* Active substance abuse, within 1 year prior to Screening
* Participation in an investigational new drug trial in the 30 days prior to Screening or within 5 half-lives of an investigational agent, whichever is longer
* Complication with malignancy Patients with a history of malignancies that have been treated with curative intent or completed chemotherapy may be eligible. Patients under evaluation for malignancy are not eligible
* Known intolerance to MRI or conditions contraindicated for MRI procedures
* Any other condition which is considered to be inappropriate for the study by the Investigator or subinvestigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in serum LDL-C at Week 16 | Week 16
  Serum

SECONDARY OUTCOMES:
Absolute change from baseline to Week 16 in the liver fat fraction (%) as measured by MRI-PDFF | Week 16
  MRI-PDFF
Absolute change from baseline to Week 16 in hepatic fibrosis as measured by MRE | Week 16
  MRE
Change from baseline to Week 16 in ALT level | Week 16
  Serum
Change from baseline to Week 16 in AST level | Week 16
  Serum
Change from baseline to Week 16 in γ-GTP level | Week 16
  Serum
Absolute change from baseline to Week 16 in HDL-C level | Week 16
  Serum
Change from baseline to Week 16 in non HDL-C level | Week 16
  Serum
Change from baseline to Week 16 in LDL-C/HDL-C ratio | Week 16
  Serum
Change from baseline to Week 16 in TG level | Week 16
  Serum

CONTACTS AND LOCATIONS:
Overall Officials: Takaomi Kessoku, MD.,PhD., Principal Investigator — Yokohama City University
Locations (1):
- Yokohama City University, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakajima A, Seki M, Taniguchi S, Ohta A, Gillberg PG, Mattsson JP, Camilleri M. Safety and efficacy of elobixibat for chronic constipation: results from a randomised, double-blind, placebo-controlled, phase 3 trial and an open-label, single-arm, phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Aug;3(8):537-547. doi: 10.1016/S2468-1253(18)30123-7. Epub 2018 May 25. PMID 29805116
- [Derived] Kessoku T, Kobayashi T, Ozaki A, Iwaki M, Honda Y, Ogawa Y, Imajo K, Saigusa Y, Yamamoto K, Yamanaka T, Usuda H, Wada K, Yoneda M, Saito S, Nakajima A. Rationale and design of a randomised, double-blind, placebo-controlled, parallel-group, investigator-initiated phase 2a study to investigate the efficacy and safety of elobixibat in combination with cholestyramine for non-alcoholic fatty liver disease. BMJ Open. 2020 Sep 9;10(9):e037961. doi: 10.1136/bmjopen-2020-037961. PMID 32907904